CLINICAL TRIAL: NCT02444728
Title: Cyclophosphamide and Hydroxychloroquine for the Treatment of Severe Thrombocytopenia in Systemic Lupus Erythematosus
Brief Title: Cyclophosphamide and Hydroxychloroquine for Thrombocytopenia in SLE
Acronym: CHORUS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Because of insufficient enrollement
Sponsor: Chinese SLE Treatment And Research Group (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTAR001
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Thrombocytopenia
Keywords: thrombocytopenia; systemic lupus erythematosus; hydroxychloroquine; cyclophosphamide; remission
MeSH Terms: conditions — Thrombocytopenia; Lupus Erythematosus, Systemic | interventions — Hydroxychloroquine; Cyclophosphamide; Azathioprine; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group1:Hydroxychloroquine (Active Comparator): Hydroxychloroquine: 100 mg tablets by mouth, 400mg everyday for 12 months Methylprednisolone: 4 mg tablets by mouth, 40-50mg everyday and tapering for 12 months
  Interventions: Drug: Hydroxychloroquine; Drug: Methylprednisolone
- Group 2:Cyclophosphamide (Active Comparator): Cyclophosphamide, Azathioprine & Methylprednisolone Cyclophosphamide: 200mg powder intravenous infusion, 1000mg every month for 6 month.
  Azathioprine: 100 mg tablets by mouth, everyday for 6 months. Methylprednisolone: 4 mg tablets by mouth, 40-50mg everyday and tapering for 12 months
  Interventions: Drug: Hydroxychloroquine; Drug: Cyclophosphamide; Drug: Azathioprine; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 200 mg BID for 12 months
  Other Names: Fenle
Drug: Cyclophosphamide — Cyclophosphamide 1000mg intravenous infusion every month for 6 months
  Other Names: Huanlinxianan
  Arms: Group 2:Cyclophosphamide
Drug: Azathioprine — After Cyclophosphamide treatment, Azathioprine 100mg once daily for 6 months
  Other Names: liuzuopiaolin
  Arms: Group 2:Cyclophosphamide
Drug: Methylprednisolone — Methylprednisolone 40-50 mg once daily for 1 months and then taped for 12 months
  Other Names: meizhuole

SUMMARY:
Treating severe thrombocytopenia is a challenge in the management of systemic lupus erythematosus. Although rheumatologists have followed some rules in real practice,there is very few evidence to support the current treatment algorithm. The purpose of this study is to compare the complete remission rate and partial remission rate of cyclophosphamide and hydroxychloroquine for treating severe thrombocytopenia in Chinese SLE patients.

DETAILED DESCRIPTION:
This is a prospective,randomized,open-label,multi-center clinical trial. The aim of this study is to test the efficacy of GC(gluco-corticosteroid)+HCQ(hydroxychloroquine) and GC(glucocorticosteroid)+CTX(cyclophosphamide) with sequential AZA(azathioprine) in the induction and maintenance therapy of severe thrombocytopenia in SLE patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients fulfilled the 1997 ACR modified or SLICC classification criteria of SLE；
2. New onset thrombocytopenia: platelet count <30X109/L(by both routine test and citric acid anti-coagulated blood count test) within 3 months

Exclusion Criteria:

1. Thrombocytopenia caused by other reasons, including drugs；
2. Positive for active HAV(hepatitis A virus)/HBV(hepatitis B virus) infection
3. Active HIV(human immunodeficiency virus) or HCV(hepatitis C virus) infection;
4. Active HP(Helicopter pylori) infection;
5. Severe liver and kidney dysfunction；
6. Severe neuropsychiatric lupus；
7. No response to high dose steroid and/or cyclophosphamide 1 month prior to study enrollment；
8. Uncontrolled diabetes or hypertension before entry
9. Active GI bleeding 3 months before entry
10. Intolerant to HCQ in the past treatment history；
11. Severe bone marrow suppression or liver damage caused by cyclophosphamide in the past history；
12. Active infection , including bacteria, virus, fungi, mycobacteria
13. Allergy to any of the study medications
14. Confirmed TTP(thrombolic thrombocytopenic purpura)or CAPS(catastrophic anti-phosphilipid syndrome)
15. Platelet count less than 20X109/L with active bleeding
16. Myelodysplastic diseases
17. Patients with heart and lung function impairment
18. thiopurine S-methyltransferase (TPMT) gene positive -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
complete remission rate | at 12 month
  percentage of patients whose platelet count > 100X109/L

SECONDARY OUTCOMES:
partial remission rate | at 12 month
  percentage of patients whose platelet increase to >30X109/L or with at least a two folds increase of the baseline(ie, pretreatment) count and the absence of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, MD, Principal Investigator — Chinese SLE Treatment And Research Group; Xiaofeng Zeng, MD, Study Chair — Peking Union Medical College Hospital; Xinping Tian, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (15):
- China (15):
  - the Affiliated Hospital to Bangbu Medical University, Bengbu, Anhui
  - Hebei Provincial Hospital, Shijiazhuang, Hebei
  - the First Affiliated Hospital of Xiangya Medical University, Changsha, Hunan
  - the Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Sino-Japanese Friendship Hospital of Jilin University, Changchun, Jilin
  - the Affiliated Hospital of Xian Communication Hospital, Xian, Shanxi
  - Xijing Hospital, Xian, Shanxi
  - Xinjiang Provincial Hospital, Ürümqi, Xinjiang
  - the Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Beijng Hospital, Beijing
  - Beijing Chaoyang Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Beijing Xuanwu Hospital, Beijing
  - General Hospital of Tianjing Medical University, Tianjin

REFERENCES:
- [Background] Abu-Shakra M, Shoenfeld Y. Azathioprine therapy for patients with systemic lupus erythematosus. Lupus. 2001;10(3):152-3. doi: 10.1191/096120301676669495. PMID 11315344
- [Background] Blasco LM. Hydroxychloroquine alone for severe immune thrombocytopenic purpura associated with systemic lupus erythematosus. Lupus. 2013 Jun;22(7):752-3. doi: 10.1177/0961203313490239. Epub 2013 May 22. No abstract available. PMID 23698017
- [Background] Cheng Y, Wong RS, Soo YO, Chui CH, Lau FY, Chan NP, Wong WS, Cheng G. Initial treatment of immune thrombocytopenic purpura with high-dose dexamethasone. N Engl J Med. 2003 Aug 28;349(9):831-6. doi: 10.1056/NEJMoa030254. PMID 12944568
- [Result] Contreras G, Tozman E, Nahar N, Metz D. Maintenance therapies for proliferative lupus nephritis: mycophenolate mofetil, azathioprine and intravenous cyclophosphamide. Lupus. 2005;14 Suppl 1:s33-8. doi: 10.1191/0961203305lu2115oa. PMID 15803929
- [Result] Neunert C, Lim W, Crowther M, Cohen A, Solberg L Jr, Crowther MA; American Society of Hematology. The American Society of Hematology 2011 evidence-based practice guideline for immune thrombocytopenia. Blood. 2011 Apr 21;117(16):4190-207. doi: 10.1182/blood-2010-08-302984. Epub 2011 Feb 16. PMID 21325604
- [Result] Boumpas DT, Barez S, Klippel JH, Balow JE. Intermittent cyclophosphamide for the treatment of autoimmune thrombocytopenia in systemic lupus erythematosus. Ann Intern Med. 1990 May 1;112(9):674-7. doi: 10.7326/0003-4819-112-9-674. PMID 2334081
- [Result] Roach BA, Hutchinson GJ. Treatment of refractory, systemic lupus erythematosus-associated thrombocytopenia with intermittent low-dose intravenous cyclophosphamide. Arthritis Rheum. 1993 May;36(5):682-4. doi: 10.1002/art.1780360516. PMID 8489547
- [Result] Levine AB, Erkan D. Clinical assessment and management of cytopenias in lupus patients. Curr Rheumatol Rep. 2011 Aug;13(4):291-9. doi: 10.1007/s11926-011-0179-5. PMID 21503695
- [Result] Khellaf M, Chabrol A, Mahevas M, Roudot-Thoraval F, Limal N, Languille L, Bierling P, Michel M, Godeau B. Hydroxychloroquine is a good second-line treatment for adults with immune thrombocytopenia and positive antinuclear antibodies. Am J Hematol. 2014 Feb;89(2):194-8. doi: 10.1002/ajh.23609. Epub 2013 Nov 20. PMID 24254965
- [Result] Arnal C, Piette JC, Leone J, Taillan B, Hachulla E, Roudot-Thoraval F, Papo T, Schaeffer A, Bierling P, Godeau B. Treatment of severe immune thrombocytopenia associated with systemic lupus erythematosus: 59 cases. J Rheumatol. 2002 Jan;29(1):75-83. PMID 11824975
- [Result] Newman K, Owlia MB, El-Hemaidi I, Akhtari M. Management of immune cytopenias in patients with systemic lupus erythematosus - Old and new. Autoimmun Rev. 2013 May;12(7):784-91. doi: 10.1016/j.autrev.2013.02.001. Epub 2013 Feb 24. PMID 23462431